CLINICAL TRIAL: NCT04663022
Title: Influence of the Sensory Profile of Deaf Children With Autism Spectrum Disorders on the Outcome of Cochlear Implantation
Acronym: PSIC-TSA
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0328
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Child with cochlear implant: 15 childs with coclear implant but without autism spectrum disorder
  Interventions: Other: Dunn's sensory profile questionnaire
- Child with cochlear implant and autism spectrum disorder: 15 childs with coclear implant and with autism spectrum disorder
  Interventions: Other: Dunn's sensory profile questionnaire

INTERVENTIONS:
Other: Dunn's sensory profile questionnaire — all children will complete the Dunn Sensory Profile questionnaire

SUMMARY:
An unpublished study conducted at Toulouse University Hospital revealed that 30% of implanted children with Autism Spectrum Disorders abandon their implant, while 70% of them keep it. The aim of this study is to evaluate the causes of this disparity, which is much greater than in children with cochlear implants without associated Autism Spectrum Disorders. Our problem is as follows: do the sensory hypersensitivity and hyposensitivity of deaf children with Autism Spectrum Disorders have an effect on the expected results after a cochlear implantation from a language and auditory reaction point of view?

DETAILED DESCRIPTION:
The present study will specifically focus on the sensory profile of these children with Autism Spectrum Disorders, which could be the cause of these developmental difficulties in language and communication development.

ELIGIBILITY:
Inclusion Criteria:

* Deaf child with cochlear implant
* 15 months to 10 years old and 6 months old at the time of implantation
* Child with autism spectrum disorder (only for children group with autisme spectrum disorder)
* No opposition from the legal representative of the authority to participate in the study

Exclusion Criteria:

* Opposition by the legal representative of the child
* Child under legal protection

Ages: 15 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population is deaf children with cochlear implant. In the first group, children must have cochlear implant and autism spectrum disorders, and in second group, children must have only cochlear implant.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
determine the sensory profile | inclusion visit
  To determine the sensory profile of implanted deaf children with autism spectrum disorders, each parent complete the questionnaire Dunn's sensory profile

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Noëlle Calmels, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France